CLINICAL TRIAL: NCT02554513
Title: Apraxia of Speech: A Comparison of EPG Treatment & Sound Production Treatment
Brief Title: Apraxia of Speech: Comparison of EPG Treatment (Tx) and Sound Production Treatment (SPT)
Acronym: EPG&SPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: C2068-P
Record Dates: First submitted 2015-08-19; First posted 2015-09-18 (Estimated); Results first posted 2021-11-04 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: Apraxia of Speech; Aphasia, Acquired; Speech Disorders
Keywords: Apraxia of Speech; Treatment
MeSH Terms: conditions — Apraxias; Aphasia; Speech Disorders

STUDY DESIGN:
Intervention Model Description: Each participant received each arm of treatment
Who Masked: Outcomes Assessor
Masking Description: Single
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EPG Tx (Active Comparator): An articulatory-kinematic treatment in conjunction with visual biofeedback specifically tongue to palate contact to improve speech production
  Interventions: Device: EPG Tx
- Sound Production Treatment (SPT) (Active Comparator): An articulatory-kinematic treatment that uses integral stimulation to improve speech production.
  Interventions: Behavioral: SPT

INTERVENTIONS:
Device: EPG Tx — behavioral intervention that incorporates a device that provides visual biofeedback
  Other Names: Electropalatography Treatment, Palatometer Treatment
  Arms: EPG Tx
Behavioral: SPT — A treatment hierarchy involving integral stimulation
  Other Names: Sound Production Treatment
  Arms: Sound Production Treatment (SPT)

SUMMARY:
The purpose of the proposed research is to examine the effects of two treatment approaches on speech production involving speakers with chronic apraxia of speech (AOS) and aphasia. The planned investigation is designed to examine the acquisition, maintenance and generalization effects of each treatment. One approach, electropalatography (EPG) uses visual biofeedback in conjunction with articulatory-kinematic treatment and the other approach, sound production treatment (SPT) is one of the most systematically studied articulatory-kinematic treatments for AOS.

DETAILED DESCRIPTION:
EPG has been used to treat apraxia of speech (AOS) as well as other speech production disorders (i.e., articulation disorders & cleft palate). SPT is one of the most systematically studied treatment approaches for AOS. Both treatment approaches are considered clinical treatment approaches/standards of care for AOS. The pseudopalate used in conjunction with EPG treatment is an acceptable device for treating speech production disorders including AOS. The pseudopalate is custom-fit for each patient and is similar to a dental retainer and is considered minimally invasive.

The purpose of this research is to systematically examine the effects of treatment on speech production using EPG treatment vs. an SPT approach. The planned investigation is intended to explicate the acquisition, maintenance, and generalization effects of each treatment approach. The specific experimental questions to be addressed are as follows:

1. Will treatment using an EPG approach or an SPT approach result in greater accuracy of articulation of trained speech sounds produced in words?
2. Will treatment using an EPG approach or an SPT approach result in greater accuracy of articulation of untrained exemplars of trained speech sounds produced in words (i.e., response generalization)?
3. Will treatment using an EPG approach or an SPT approach result in greater long term maintenance effects for trained speech sounds?
4. Do different treatment approaches result in distinct ratings of functional communication skills via the Aphasia Communication Outcome Measure (ACOM; Doyle et al., 2012) and an outcome measure of speech intelligibility using the Assessment of Intelligibility of Dysarthric Speech (AIDS; Yorkston & Beukelman, 1981)?

ELIGIBILITY:
Inclusion Criteria:

* Veterans or non Veterans with apraxia of speech who reside in the Salt Lake City region (commutable),
* 6 months or more post stroke or other focal brain injury, no other neurological conditions
* native English speakers, hearing adequate for experimental task (e.g., pass puretone screening at 35dB at 500, 1K, 2K Hz or adequate aided hearing)
* non linguistic cognition within normal limits

Exclusion Criteria:

* less than 6 months post stroke
* insufficient hearing, insufficient non linguistic cognitive skills
* neurological conditions other than stroke
* unable to attend treatment in the Salt Lake City vicinity

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-11-02 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shannon C Mauszycki, PhD, Principal Investigator — VA Salt Lake City Health Care System, Salt Lake City, UT
Locations (1):
- VA Salt Lake City Health Care System, Salt Lake City, UT, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mauszycki SC, Wambaugh JL. Acquired Apraxia of Speech: Comparison of Electropalatography Treatment and Sound Production Treatment. Am J Speech Lang Pathol. 2020 Feb 21;29(1S):511-529. doi: 10.1044/2019_AJSLP-CAC48-18-0223. Epub 2019 Nov 6. PMID 31693389

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Each participant received each treatment arm in this crossover design. Order of treatment assignment was random.
Groups:
- EPG Tx Then Sound Production Treatment (SPT): Participants in this arm received EPG Treatment for 20 treatment sessions. Following a 2 week washout period, participants received Sound Production Treatment (SPT) for 20 treatment sessions.
  EPG Treatment is also a behavioral treatment that includes clinical modeling, integral stimulation ("watch me, listen to me, say it with me"), articulation instruction, repeated practice and verbal feedback, but also incorporates a device that provides visual feedback about tongue placement/movements for articulation.
  SPT is a behavioral treatment that includes clinician modeling, orthographic cueing, integral stimulation ("watch me, listen to me, say it with me"), articulation instruction, repeated practice and verbal feedback.
- Sound Production Treatment (SPT) Then EPG Tx: Participants in this arm received Sound Production Treatment - Blocked (SPT) for 20 treatment sessions. Following a 2 week washout period, participants received EPG Treatment for 20 treatment sessions.
  SPT is a behavioral treatment that includes clinician modeling, orthographic cueing, integral stimulation ("watch me, listen to me, say it with me"), articulation instruction, repeated practice and verbal feedback.
  EPG Treatment is also a behavioral treatment that includes clinical modeling, integral stimulation ("watch me, listen to me, say it with me"), articulation instruction, repeated practice and verbal feedback, but also incorporates a device that provides visual feedback about tongue placement/movements for articulation.
Period: First Treatment Phase (7 Weeks)
Arm/Group | EPG Tx Then Sound Production Treatment (SPT) | Sound Production Treatment (SPT) Then EPG Tx
Started | 3 | 3
Completed | 3 | 2
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Washout (2 Weeks)
Arm/Group | EPG Tx Then Sound Production Treatment (SPT) | Sound Production Treatment (SPT) Then EPG Tx
Started | 3 | 2
Completed | 3 | 2
Not Completed | 0 | 0
Period: Second Treatment Phase (7 Weeks)
Arm/Group | EPG Tx Then Sound Production Treatment (SPT) | Sound Production Treatment (SPT) Then EPG Tx
Started | 3 | 2
Completed | 3 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants had moderate to severe acquired apraxia of speech and accompanying aphasia.
Groups:
- All Participants: All participants received Electropalatography Treatment (EPG Tx) and Sound Production Treatment (SPT). Half the participants received EPG Tx first for 20 sessions. Following a 2 week washout period, those participants then received SPT for 20 sessions. The other half of the participants received the treatments in the opposite order.
Arm/Group | All Participants
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.6 (15.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Speech Production: Percent Change in Treated Items Immediately Post Treatment
Description: Change in accuracy of articulation of treated items measured by percent increase in accuracy above the highest baseline measurement; production of words designated for treatment was measured repeatedly in non-treatment probes prior to treatment, throughout all study phases and immediately post treatment with percent accuracy calculated for each probe (0% to 100% correct). The highest percentage accuracy achieved in baseline probes was subtracted from the percentage accuracy achieved at the conclusion of treatment to obtain change in accuracy value - this reflects change from maximum correct performance in baseline (baseline). e.g., if in baseline probes, performance ranged from 10% to 30% accuracy and at post treatment performance was 90% accuracy, the change value would be 60% (90% minus 30%). A greater value indicates greater change in articulation/production of words. Change could be positive (improved articulation) or negative (poorer articulation)
Time Frame: Baseline vs. Immediately Post Treatment (7 week treatment period)
Measure: Mean (Full Range); unit: % change
Groups:
- EPG Treatment: EPG Treatment: Articulatory-Kinematic Treatment in conjunction with visual biofeedback for tongue position
- Sound Production Treatment: Sound Production Treatment: Articulatory-Kinematic Treatment
Arm/Group | EPG Treatment | Sound Production Treatment
Number analyzed (Participants) | 5 | 5
% change | 59 [40 to 78] | 66 [62 to 70]

2. Secondary Outcome: Speech Production: Percent Change in Untreated Items (Related Items) Immediately Post Treatment
Description: Change in articulatory accuracy of untreated items, but related items as measured by percent increase in accuracy above the highest baseline measurement; production of words designated for non-treatment was measured repeatedly in non-treatment probes prior to treatment, throughout all study phases and immediately post treatment with percent accuracy calculated for each probe (0% to 100% correct). The highest percentage accuracy achieved in baseline probes was subtracted from the percentage accuracy achieved at the conclusion of treatment to obtain change in accuracy value - this reflects change from maximum correct performance in baseline. e.g., if in baseline probes, performance ranged from 10% to 30% accuracy and at post treatment performance was 90% accuracy, the change value would be 60% (90% minus 30%). A greater change value indicates greater change in articulation/production of words. Change could be positive (improved articulation) or negative (poorer articulation)
Time Frame: Baseline vs. Immediately Post Treatment (7 week treatment period)
Measure: Mean (Full Range); unit: % change
Groups:
- Treatment With EPG: Participants received articulatory-kinematic treatment in conjunction with visual-biofeedback via electropalatography (i.e., tongue movement/placement)
- Sound Production Treatment: Participants received articulatory-kinematic treatment
Arm/Group | Treatment With EPG | Sound Production Treatment
Number analyzed (Participants) | 5 | 5
% change | 5 [0 to 10] | 50 [40 to 60]

3. Secondary Outcome: Speech Production: Percent Change for Treated Items After the Completion of Treatment
Description: Change in articulatory accuracy of treated items as measured by percent increase in accuracy above the highest baseline measurement; production of words designated for treatment was measured repeatedly in non-treatment probes prior to treatment, throughout all study phases, and at 7 weeks immediately after each treatment with percent accuracy calculated for each probe (0% to 100% correct). The highest percentage accuracy achieved in baseline probes was subtracted from the percentage accuracy achieved at 7 weeks immediately after the conclusion of each treatment to obtain change in accuracy value - this reflects change from maximum correct performance in baseline (pre-treatment). e.g., if in baseline probes, performance ranged from 10% to 30% accuracy and at post treatment performance was 90% accuracy, the change value would be 60% (90% minus 30%). A greater change value indicates greater change in articulation/production of words.
Time Frame: Baseline vs. 7 weeks post treatment [measured immediately after the completion of each treatment]
Measure: Mean (Full Range); unit: % change
Groups:
- Treatment With EPG: An articulatory-kinematic treatment in conjunction with visual biofeedback for tongue position
- Sound Production Treatment: An articulatory-kinematic treatment
Arm/Group | Treatment With EPG | Sound Production Treatment
Number analyzed (Participants) | 5 | 5
% change | 43 [20 to 66] | 61 [45 to 77]

4. Secondary Outcome: Functional Communication Skills: T-Score
Description: Measurement of functional every day communication skills using the Aphasia Communication Outcome Measure (ACOM) with a T-score computed at each administration which was at baseline and then 10 weeks after the completion of all treatment. This outcome measure was only completed at baseline and at the completion on all treatment [not measured after the completion of each treatment]. The rating scale for functional communication skills was completed by the patient (or a spouse if patient's auditory comprehension was significantly impaired) (T-Scores range from 0 to 100; Higher T-scores indicate greater functional communication skills)
Time Frame: Baseline vs. 10 weeks after the completion of all treatment [measured at pre-treatment and post-treatment; conclusion of all treatment]
Measure: Mean (Standard Deviation); unit: T-Score
Groups:
- All Participants - Pre vs. Post Treatment: Aphasia Communication Outcome Measure (ACOM)
Arm/Group | All Participants - Pre vs. Post Treatment
Number analyzed (Participants) | 5
T-Score
  Pre-Treatment | 43.0 (16)
  Post-Treatment | 46.0 (21)

5. Secondary Outcome: Speech Intelligibility: Percentage
Description: Measurement of speech intelligibility for a set of fifty words (non-treatment words) from the Assessment of Speech Intelligibility of Dysarthric Speech as judge by an unfamiliar listener that was measured at baseline and then at 10 weeks post all treatment with a percentage of speech intelligibility (0% to 100% intelligible).This measurement was only conducted at pre-treatment and at the conclusion of all treatment [not measured after each treatment].
Time Frame: Baseline vs. 10 weeks post all treatment [measured at pre-treatment and post-treatment; conclusion of all treatment]
Measure: Mean (Standard Deviation); unit: Percentage of Words Intelligible
Groups:
- All Participants - Pre vs. Post Treatment: Assessment of Intelligibility of Dysarthric Speech (ASSIDS) - Word Level
Arm/Group | All Participants - Pre vs. Post Treatment
Number analyzed (Participants) | 5
Percentage of Words Intelligible
  Pre-Treatment | 40.0 (30)
  Post-Treatment | 50.0 (25)

ADVERSE EVENTS:
Time Frame: Entire course of study which was approximately 32 weeks per participant: pretreatment/baseline period = 6 weeks + 7 weeks Treatment 1 + 2 weeks washout + 7 weeks Treatment 2 + follow-up at 10 weeks.
Groups:
- EPG Treatment: All Participants: Participants in this arm received EPG Treatment for 20 treatment sessions. Following a 2 week washout period, participants received Sound Production Treatment (SPT) for 20 treatment sessions.
  EPG Treatment is also a behavioral treatment that includes clinical modeling, integral stimulation ("watch me, listen to me, say it with me"), articulation instruction, repeated practice and verbal feedback, but also incorporates a device that provides visual feedback about tongue placement/movements for articulation.
  SPT is a behavioral treatment that includes clinician modeling, orthographic cueing, integral stimulation ("watch me, listen to me, say it with me"), articulation instruction, repeated practice and verbal feedback.
- Sound Production Treatment: All Participants: Participants in this arm received Sound Production Treatment - Blocked (SPT) for 20 treatment sessions. Following a 2 week washout period, participants received EPG Treatment for 20 treatment sessions.
  SPT is a behavioral treatment that includes clinician modeling, orthographic cueing, integral stimulation ("watch me, listen to me, say it with me"), articulation instruction, repeated practice and verbal feedback.
  EPG Treatment is also a behavioral treatment that includes clinical modeling, integral stimulation ("watch me, listen to me, say it with me"), articulation instruction, repeated practice and verbal feedback, but also incorporates a device that provides visual feedback about tongue placement/movements for articulation.
Arm/Group | EPG Treatment: All Participants | Sound Production Treatment: All Participants
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-12): https://cdn.clinicaltrials.gov/large-docs/13/NCT02554513/Prot_SAP_000.pdf